CLINICAL TRIAL: NCT05678803
Title: Short-Term Outcomes Of Subaxial Cervical Injuries in Assiut University Trauma Center
Brief Title: Short-Term Outcomes Of Subaxial Cervical Injuries
Status: Completed | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Peter Nabil Gayed Abdelmalak, Principal investigator, Assiut University
Other Study IDs: Subaxial Cervical Injuries
Record Dates: First submitted 2022-02-09; First posted 2023-01-10 (Actual); Last update posted 2023-05-10 (Actual); Status verified 2023-05

CONDITIONS: Cervical Spinal Cord Injury
MeSH Terms: interventions — X-Rays

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: xrays and CT — A dedicated sheet will be used to record patients' data including all demographic data, detailed analysis of the mechanism of injury, time of injury, time and details of surgery (if any), neurological status on admission and all radiological findings. All patients will undergo plain X-rays and CT imaging. Patients with suspected discoligamentous injuries and/or neurological deficits will also be assessed by MRI.

SUMMARY:
The subaxial cervical spine consists of levels C3 through C7 and includes both the bony anatomy as well as the ligamentous anatomy. Injuries to the subaxial cervical spine can be bony, discoligamentous or a combination of both (1). Cervical spine trauma is common resulting from high energy trauma such as falling from height and motor vehicle accident (2). Devastating sequelae of subaxial cervical spine trauma include quadriplegia, functional loss, and permanent disability

DETAILED DESCRIPTION:
Initially, all patients with subaxial cervical spine fractures require immobilization in a rigid cervical orthosis (2). Patients receiving conservative treatment are often prescribed a rigid cervical or cervicothoracic orthosis for 6 to 12 weeks with regular follow-up and interval radiographs to assess alignment.

Patients with fractures deemed unstable or neurologic compromise should undergo decompression and stabilization. Intervention within 24 hours of injury leads to better improvement in ASIA scores (3). The recent AO Spine Subaxial Classification system relies essentially on MSCT evaluation (Reference). However, MRI is superior to CT scans for evaluating the spinal cord, nerve roots, disc, and ligamentous structures in the cervical spine (4).

Even though the investigators receive and treat a large number of patients with various subaxial cervical injuries in Assiut University Hospital each year, there is no consensus about the best treatment options and uncertainty about the outcome of these treatments.

In this study, the participants will assess the short-term outcomes of all patients with subaxial cervical fractures who will be admitted to the participants' center regardless of the neurological status or treatment type used.

The participants will also create a detailed prospective database to be used for another later study on the long-term outcome

ELIGIBILITY:
Inclusion Criteria:

* All patients presenting with subaxial cervical spine injuries with and without cervical cord injury between January 2022 and December 2022.

Exclusion Criteria:

* 1- Patients who refuse to participate in the study 2- Patients who are not available for 6 weeks follow up

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients presenting with subaxial cervical spine injuries with and without cervical cord injury between January 2022 and December 2022.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2022-03-10 (Actual); Primary Completion 2023-03-09 (Actual); Study Completion 2023-03-09 (Actual)

PRIMARY OUTCOMES:
Short-Term Outcomes Of Subaxial Cervical Injuries in Assiut University Trauma Center | 1 year
  Neck disability index It is a standard instrument for measuring self-rated disability due to neck pain and is used by both clinicians and researchers. Each of the 10 items scores from 0 to 5. The maximum score is 50. The obtained score can be multiplied by two to produce a percentage score

CONTACTS AND LOCATIONS:
Locations (1):
- Peternabil049@Gmail.Com, Asyut, Egypt

REFERENCES:
- [Background] Stauffer ES. Subaxial injuries. Clin Orthop Relat Res. 1989 Feb;(239):30-9. PMID 2912631
- [Background] Feuchtbaum E, Buchowski J, Zebala L. Subaxial cervical spine trauma. Curr Rev Musculoskelet Med. 2016 Dec;9(4):496-504. doi: 10.1007/s12178-016-9377-0. PMID 27864669
- [Background] Schroeder GD, Vaccaro AR. Cervical Spine Injuries in the Athlete. J Am Acad Orthop Surg. 2016 Sep;24(9):e122-33. doi: 10.5435/JAAOS-D-15-00716. PMID 27479833
- [Background] Kwon BK, Vaccaro AR, Grauer JN, Fisher CG, Dvorak MF. Subaxial cervical spine trauma. J Am Acad Orthop Surg. 2006 Feb;14(2):78-89. doi: 10.5435/00124635-200602000-00003. PMID 16467183
- [Background] Pourtaheri S, Emami A, Sinha K, Faloon M, Hwang K, Shafa E, Holmes L Jr. The role of magnetic resonance imaging in acute cervical spine fractures. Spine J. 2014 Nov 1;14(11):2546-53. doi: 10.1016/j.spinee.2013.10.052. Epub 2013 Nov 22. PMID 24269913
- [Background] Shaheen AA, Omar MT, Vernon H. Cross-cultural adaptation, reliability, and validity of the Arabic version of neck disability index in patients with neck pain. Spine (Phila Pa 1976). 2013 May 1;38(10):E609-15. doi: 10.1097/BRS.0b013e31828b2d09. PMID 23429690